CLINICAL TRIAL: NCT06254040
Title: Randomized, Triple-blind, Parallel-group Study to Evaluate the Effect of Consuming a Mixture of Extracts and DHA on the Mild Cognitive Impairment
Brief Title: Effect of Consuming a Mixture of Extracts and DHA on the Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C029
Record Dates: First submitted 2022-08-24; First posted 2024-02-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment
Keywords: DHA; plant extracts; cognitive; brain
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Volunteers will take 1 dissolving powder pack with maltodextrin daily for 6 months.
  Interventions: Dietary Supplement: Placebo
- Experimental Group (Experimental): Volunteers will take 1 dissolving powder pack with the mixture of extracts and DHA daily for 6 months.
  Interventions: Dietary Supplement: mixture of extracts and DHA

INTERVENTIONS:
Dietary Supplement: Placebo — Each participant will consume 1 dissolving powder pack per day diluted in water, with breakfast, without any restriction in the diet or in their life habits.
  Arms: Control Group
Dietary Supplement: mixture of extracts and DHA — Each participant will consume 1 dissolving powder pack per day diluted in water, with breakfast, without any restriction in the diet or in their life habits.
  Arms: Experimental Group

SUMMARY:
The objective of this trial is to evaluate the effect of the consumption of a mixture of extracts and DHA on the mild cognitive impairment.

DETAILED DESCRIPTION:
According to the World Health Organization, around 50 million people in the world have dementia, so developing new strategies to prevent cognitive impairment is an important aspect.

Certain plant extracts have properties related to the improvement of brain function. In addition, adequate levels of DHA are essential for good cognitive functioning throughout the life cycle.

Therefore, the objective of this trial is to evaluate the effect of the consumption of a mixture of extracts and DHA on the mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 50 years of age at the time of the screening visit.
* Mild cognitive impairment according to multidomain criteria.
* Mini Mental State Examination (MMSE) ≥21.
* Availability of an accompanying who is responsible for the patient taking the study product and attending visits.
* Patients and accompanying who agree to sign the informed consent before performing any study procedure and after they have been informed about the methods and limitations of the study.

Exclusion Criteria:

* Inability to perform neurocognitive tests.
* Intake currently (or in the two weeks prior to the start the study) of nutraceuticals that may alter the results of the study: vitamin complexes, omega-3 supplements, omega-3 fortified foods, ginkgo supplements, or any other specific supplement for memory improvement.
* Consumption of anti-dementia drugs such as memantine or cholinesterase inhibitors (ICE).
* Consumption of benzodiazepines in unstable doses.
* Severe psychiatric pathology.
* Allergy to any of the ingredients of the study product or placebo (lactose intolerance, intolerance to milk protein or allergy to any of the extracts used).

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Score of the Delayed Memory test. | 6 months
  Wechsler Memory Scale III questionnaire, delayed recall

SECONDARY OUTCOMES:
Score of the Mini Mental State Examination test. | 6 months
  Total score obtained in tests of: orientation, fixation, calculation and attention, memory, language and construction.
Score of the Immediate Memory test. | 6 months
  Wechsler Memory Scale III questionnaire, immediate recall.
Total score of the ADAS-cog neurocognitive test. | 6 months
  Total score obtained in tests of: word recall, commands, object and finger naming, constructive praxis, ideational praxis, orientation, word recognition, memory test instruction recall, spoken language ability, spoken language comprehension, difficulty finding the right words.
Analysis of plasma levels of interleukins IL-6 to inflammatory parameters. | 6 months
  Levels of interleukins IL-6
Analysis of plasma levels of interleukins IL-2 to inflammatory parameters. | 6 months
  Levels of interleukins IL-2
Analysis of plasma levels of interleukins IL-10 to inflammatory parameters. | 6 months
  Levels of interleukins IL-10
Analysis of plasma levels of PTX3 to inflammatory parameters. | 6 months
  Levels of PTX3
Analysis of plasma levels of SAP to inflammatory parameters. | 6 months
  Levels of SAP.
Analysis of plasma levels of glucose related to glucose metabolism. | 6 months
  Levels of glucose
Analysis of plasma levels of insulin related to glucose metabolism. | 6 months
  Levels of insulin
Index of the HOMA IR | 6 months
  Index of the HOMA IR

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Blanco Rojo, PhD, Principal Investigator — Biosearch S.A.
Locations (1):
- Complejo hospitalario Ruber Juan Bravo. Servicio de Neurología y Neurofisiología, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No